CLINICAL TRIAL: NCT01850524
Title: A Phase 3, Randomized, Double-Blind, Multicenter Study Comparing Oral MLN9708 Plus Lenalidomide and Dexamethasone Versus Placebo Plus Lenalidomide and Dexamethasone in Adult Patients With Newly Diagnosed Multiple Myeloma
Brief Title: IXAZOMIB Plus Lenalidomide and Dexamethasone Versus Placebo Plus Lenalidomide and Dexamethasone in Adult Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C16014; 2013-000326-54 (EudraCT Number); U1111-1158-2646 (Registry Identifier: WHO); 163325 (Registry Identifier: HC-CTD)
Record Dates: First submitted 2013-04-26; First posted 2013-05-09 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed multiple myeloma; multiple myeloma; MLN9708; IXAZOMIB; Proteasome inhibitor; Tourmaline MM2
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Dexamethasone; Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + LenDex (Placebo Comparator): Participants who were randomly assigned to receive placebo matching capsule single oral dose on Days 1, 8 and 15 along with standard regimen of LenDex (lenalidomide 25 mg capsules orally on Days 1-21 and dexamethasone 40 mg tablets orally on Days 1, 8, 15 and 22) for the first 18 cycles (each cycle was of 28 days). Following Cycle 18, participants received 3.0 mg ixazomib matching placebo capsule as single oral dose on Days 1, 8 and 15 along with lenalidomide 10 mg capsules orally on Days 1-21 in each 28-day cycle until progressive disease or unacceptable toxicity, whichever comes first up to end of study (up to approximately 109 months).
  Interventions: Drug: Placebo; Drug: Dexamethasone; Drug: Lenalidomide
- Active Comparator: Ixazomib + LenDex (Active Comparator): Participants who were randomly assigned to receive Ixazomib 4.0 mg capsule single oral dose on Days 1, 8 and 15 along with standard regimen of LenDex (lenalidomide 25 mg capsules orally on Days 1-21 and dexamethasone 40 mg tablets orally on Days 1, 8, 15 and 22) for the first 18 cycles (each cycle was of 28 days). Following Cycle 18, participants received 3.0 mg ixazomib capsule as single oral dose on Days 1, 8 and 15 along with lenalidomide 10 mg capsules orally on Days 1-21 in each 28-day cycle until progressive disease or unacceptable toxicity, whichever comes first up to end of study (up to approximately 109 months).
  Interventions: Drug: Ixazomib; Drug: Dexamethasone; Drug: Lenalidomide

INTERVENTIONS:
Drug: Ixazomib — IXAZOMIB capsules.
  Other Names: MLN9708
  Arms: Active Comparator: Ixazomib + LenDex
Drug: Placebo — IXAZOMIB matching-placebo capsules.
  Arms: Placebo + LenDex
Drug: Dexamethasone — Dexamethasone tablets.
Drug: Lenalidomide — Lenalidomide capsules.

SUMMARY:
The purpose of this study is to provide continued access to ixazomib and/or lenalidomide to participants who are continuing to have clinical benefit and to continue collecting relevant safety data to monitor safety in participants with Newly Diagnosed Multiple Myeloma (NDMM) who are not eligible for stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years or older diagnosed with Multiple Myeloma according to standard criteria who have not received prior treatment for multiple myeloma.
2. Participants for whom lenalidomide and dexamethasone treatment is appropriate and who are not eligible for high-dose therapy followed by stem-cell transplantation (HDT-SCT) for 1 or more of the following reasons:

   * The participant is 65 years of age or older.
   * The participant is less than 65 years of age but has significant comorbid condition(s) that are, in the opinion of the investigator, likely to have a negative impact on tolerability of HDT-SCT.
3. Measurable disease as specified in study protocol.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. Meet the clinical laboratories criteria as specified in the protocol.
6. Female participants who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or agree to practice true abstinence, and must also agree to ongoing pregnancy testing; must also adhere to the guidelines of the lenalidomide pregnancy prevention program.
7. Male participants who agree to practice effective barrier contraception or agree to practice true abstinence AND must adhere to the guidelines of the lenalidomide pregnancy prevention program.
8. Suitable venous access for the study-required blood sampling.
9. Must be able to take concurrent aspirin 70 mg to 325 mg daily (or enoxaparin if aspirin allergic).
10. Voluntary written consent.
11. Participant is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Prior treatment for multiple myeloma with either standard of care treatment or investigational regimen.
2. Diagnosed and treated for another malignancy within 5 years before randomization or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
3. Inability or unwillingness to receive antithrombotic therapy.
4. Female participants who are lactating or pregnant.
5. Major surgery or radiotherapy within 14 days before randomization.
6. Infection requiring intravenous antibiotics within 14 days before the first dose of study drug.
7. Central nervous system involvement.
8. Diagnosis of Waldenstrom's macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome, plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome.
9. Evidence of current uncontrolled cardiovascular conditions within 6 months prior to randomization, including: Uncontrolled hypertension, cardiac arrhythmias, or congestive heart failure; Unstable angina, or Myocardial infarction.
10. Systemic treatment with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin,itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort within 14 days before randomization in the study.
11. Active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
12. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the participant inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens (e.g., peripheral neuropathy that is Grade 1 with pain or Grade 2 or higher of any cause).
13. Psychiatric illness/social situation that would limit compliance with study requirements.
14. Known allergy to any of the study medications.
15. Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or gastrointestinal (GI) procedure that could interfere with the oral absorption or tolerance of treatment.
16. Treatment with any investigational products within 60 days before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2013-04-29 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2022-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (147):
- United States (78):
  - Birmingham, Alabama
  - Chandler, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Corona, California
  - Fountain Valley, California
  - Fullerton, California
  - Irvine, California
  - La Jolla, California
  - Mission Hills, California
  - Oakland, California
  - Riverside, California
  - San Diego, California
  - San Jose, California
  - San Leandro, California
  - Santa Clara, California
  - South San Francisco, California
  - Vallejo, California
  - Denver, Colorado
  - Fort Collins, Colorado
  - Hartford, Connecticut
  - Plainville, Connecticut
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Honolulu, Hawaii
  - Iowa City, Iowa
  - Sioux City, Iowa
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Towson, Maryland
  - Burlington, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Lansing, Michigan
  - Southfield, Michigan
  - Duluth, Minnesota
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Bridgeton, Missouri
  - Kansas City, Missouri
  - Little Silver, New Jersey
  - Albuquerque, New Mexico
  - Farmington, New Mexico
  - Las Cruces, New Mexico
  - Buffalo, New York
  - Lake Success, New York
  - New York, New York
  - Poughkeepsie, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Scranton, Pennsylvania
  - Charleston, South Carolina
  - Cookeville, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Galveston, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Tyler, Texas
  - Christiansburg, Virginia
  - Richmond, Virginia
  - Everett, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Vancouver, Washington
  - Yakima, Washington
- Belgium (7):
  - Brussels, Brussels Capital
  - Yvoir, Namur
  - Ghent, Oost-Vlaanderen
  - Leuven, Vlaams Brabant
  - Roeselare, West-Vlaanderen
  - Bruges
  - Liège
- Canada (12):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Surrey, British Columbia
  - Victoria, British Columbia
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Fleurimont, Quebec
  - Lévis, Quebec
  - Montreal, Quebec
- France (37):
  - Nice, Alpes-Maritimes
  - Strasbourg, Bas-Rhin
  - Brest, Finistere
  - Saint-Brieuc, Finistere
  - Limoges, Haute-Vienne
  - Castelnau-le-Lez, Herault
  - La Tronche, Isere
  - Nantes, Loire-Atlantique
  - Angers, Maine-et-Loire
  - Reims, Marne
  - Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Vannes, Morbihan
  - Lille, Nord
  - Lens, Pas-de-Calais
  - Saint-Priest-en-Jarez, Rhone
  - Montivilliers, Seine-Maritime
  - Poitiers, Vienne
  - Amiens
  - Bayonne
  - Bordeaux
  - Caen
  - Chalon-sur-Saône
  - Créteil
  - Dunkirk
  - La Roche-sur-Yon
  - Le Chesnay
  - Le Mans
  - Lille
  - Montpellier
  - Mulhouse
  - Paris
  - Périgueux
  - Pierre-Bénite
  - Pontoise
  - Rouen
  - Toulouse
  - Tours
- New Zealand (5):
  - Auckland, North Island
  - Wellington, North Island
  - Christchurch, South Island
  - Dunedin, South Island
  - Hamilton
- Ryazan, Russia
- South Korea (7):
  - Goyang, Gyeonggido
  - Seongnam-si, Gyeonggido
  - Daegu
  - Daejeon
  - Incheon
  - Jeongnam
  - Seoul

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Facon T, Venner CP, Bahlis NJ, Offner F, White DJ, Karlin L, Benboubker L, Rigaudeau S, Rodon P, Voog E, Yoon SS, Suzuki K, Shibayama H, Zhang X, Twumasi-Ankrah P, Yung G, Rifkin RM, Moreau P, Lonial S, Kumar SK, Richardson PG, Rajkumar SV. Oral ixazomib, lenalidomide, and dexamethasone for transplant-ineligible patients with newly diagnosed multiple myeloma. Blood. 2021 Jul 1;137(26):3616-3628. doi: 10.1182/blood.2020008787. PMID 33763699
- See also: Related Info — https://www.tourmalinetrialmm2.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 238 investigative sites in multiple countries from 29 April 2013 to 24 June 2022.
Pre-assignment Details: Participants with newly diagnosed multiple myeloma were enrolled in 1:1 ratio to receive ixazomib or placebo in addition to the background therapy of Lenalidomide and Dexamethasone (LenDex) in this study.
Groups:
- Ixazomib + LenDex: Participants who were randomly assigned to receive Ixazomib 4.0 mg capsule single oral dose on Days 1, 8 and 15 along with standard regimen of LenDex (lenalidomide 25 mg capsules orally on Days 1-21 and dexamethasone 40 mg tablets orally on Days 1, 8, 15 and 22) for the first 18 cycles (each cycle was of 28 days). Following Cycle 18, participants received 3.0 mg ixazomib capsule as single oral dose on Days 1, 8 and 15 along with lenalidomide 10 mg capsules orally on Days 1-21 in each 28-day cycle until progressive disease or unacceptable toxicity, whichever comes first up to end of study (up to approximately 109 months).
Period: Overall Study
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Started | 354 | 351
Intent-to-Treat (ITT) Population | 354 | 351
Safety Population (Includes all treated participants. Participants were analyzed as treated.) | 349 (1 participant in this arm who withdrew from the study was not included in the safety population.) | 354 (Included 4 participants from placebo who received ixazomib; 1 participant who withdrew was excluded.)
Participants Completed Study Treatment Per Protocol (Includes participants who completed treatment per protocol until disease progression or until discontinuation for unacceptable toxicity, withdrawal of consent, or death.) | 283 | 284
Per Protocol (PP) Population | 293 | 296
Participants With Exposure of ≥ 19 Cycles | 189 | 191
Response-evaluable Population (Includes all participants in the ITT population who receive at least 1 dose of any study drug, have measurable disease at baseline, and at least 1 post baseline response assessment assessed by an Independent Review Committee (IRC).) | 347 | 335
Completed (Completed=who completed the study.) | 183 | 178
Not Completed | 171 | 173
Not completed — Lost to Follow-up | 5 | 10
Not completed — Withdrawal by Subject | 24 | 22
Not completed — Reason not Specified | 142 | 141

BASELINE CHARACTERISTICS:
Population: ITT population included all participants who are randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + LenDex | Ixazomib + LenDex | Total
Number analyzed (Participants) | 354 | 351 | 705
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (5.91) | 73.5 (6.53) | 73.6 (6.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 179 | 351
  Male | 182 | 172 | 354
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 12 | 26
  Not Hispanic or Latino | 340 | 337 | 677
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 52 | 44 | 96
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 13 | 11 | 24
  White | 285 | 291 | 576
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  France | 136 | 126 | 262
  Belgium | 37 | 36 | 73
  Russia | 3 | 2 | 5
  Japan | 28 | 31 | 59
  South Korea | 20 | 11 | 31
  New Zealand | 3 | 3 | 6
  United States | 68 | 79 | 147
  Canada | 59 | 63 | 122
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed indicates number of participants available for analysis at baseline.
  cm
    number analyzed (Participants) | 341 | 339 | 680
    (all) | 164.7 (10.04) | 164.3 (10.13) | 164.5 (10.08)
Weight [Mean (Standard Deviation); unit: kg] | 70.53 (15.353) | 72.67 (16.995) | 71.59 (16.215)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — BSA = square root of (height x weight/3600) Population: Number analyzed indicates number of participants available for analysis at baseline.
  m^2
    number analyzed (Participants) | 341 | 339 | 680
    (all) | 1.789 (0.2306) | 1.810 (0.2456) | 1.800 (0.2383)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of first documentation of progressive disease (PD) or death due to any cause according to International Myeloma Working Group (IMWG) criteria whichever occurs first. PD required one of the following: Increase of >=25% from nadir in: Serum M-component and/or (the absolute increase must be >=0.5 g/dL); Urine M-component and/or (the absolute increase must be >=200 mg/24 hours); in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain (FLC) levels (absolute increase must be > 10 mg/dL); Bone marrow plasma cell percentage: the absolute % must be >10%; development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; hypercalcemia (corrected serum calcium > 11.5 mg/dL or 2.85 mmol/L).
Time Frame: Up to approximately 79 months
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 354 | 351
months | 21.8 [19.65 to 30.78] | 35.3 [26.45 to 43.70]
Statistical Analysis 1: Comparison: Placebo + LenDex vs Ixazomib + LenDex; Test type: Superiority; p = 0.073, Log Rank; Log-rank test is stratified by age (<75 years vs >=75), ISS (stage I or II vs stage III), and BPI-SF worst pain score (<4 vs >=4) at screening; Hazard Ratio (HR) = 0.830, 95% CI 2-sided [0.676 to 1.018]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death. Participants without documented death at the time of analysis are censored at the date last known to be alive.
Time Frame: From the date of randomization to death due to any cause (Up to approximately 9 years)
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 354 | 351
months | NA [58.71 to NA] — Median and Upper limit of Confidence Interval (CI) was not estimable due to censoring of participants as most participants were still alive during last contact. | NA [63.18 to NA] — Median and Upper limit of CI was not estimable due to censoring of participants as most participants were still alive during last contact.
Statistical Analysis 1: Comparison: Placebo + LenDex vs Ixazomib + LenDex; Test type: Superiority; p = 0.988, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.998, 95% CI 2-sided [0.790 to 1.261] — Hazard ratio is based on an Unadjusted Cox's proportional hazard regression model is stratified by age (<75 years vs >=75), ISS (stage I or II vs stage III), and BPI-SF worst pain score (<4 vs >=4) at screening

3. Secondary Outcome: Complete Response (CR) Rate
Description: CR rate was defined as the percentage of participants who achieve CR assessed by an IRC relative to the intent-to-treat (ITT) population during the treatment period. Percentage of participants with CR, as assessed by IMWG disease assessment criteria were reported. CR was defined as negative immunofixation of serum and urine along with the disappearance of any soft tissue plasmacytomas and <5 % plasma cells (PC's) in bone marrow.
Time Frame: Up to approximately 9 years
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 354 | 351
percentage of participants | 14 | 26
Statistical Analysis 1: Comparison: Placebo + LenDex vs Ixazomib + LenDex; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; CMH test is stratified by age (<75 years vs >=75), ISS (stage I or II vs stage III), and BPI-SF worst pain score (<4 vs >=4) at screening; Odds Ratio (OR) = 2.10, 95% CI 2-sided [1.43 to 3.09] — Odds ratio and confidence interval are based on logistic regression model with treatment group as categorical predictor variable,age(<75 years vs >=75), ISS(stage I or II vs stage III),and BPI-SF worst pain score(<4 vs >=4)at screening as covariates

4. Secondary Outcome: Pain Response Rate as Assessed by the Brief Pain Inventory- Short Form (BPI-SF) and Analgesic Use
Description: Pain response rate was defined as percentage of participants with pain response. Pain response was defined as the occurrence of at least a 30% reduction from baseline in BPI-SF worst pain score over the last 24 hours without an increase in analgesic use for 2 consecutive measurements > 28 days apart, were reported. Brief Pain Inventory - Short Form (m-BPI-SF) is a participant rated 11-point Likert rating scale ranged from 0 (no pain) to 10 (worst pain imaginable). Percentages are rounded off to the nearest single decimal.
Time Frame: Up to approximately 9 years
Population: ITT population included all participants who were randomized. Overall number of participants analyzed are the number of participants with baseline worst pain score>=4 as assessed by m-BPI-SF.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 195 | 190
percentage of participants | 51.3 | 50.5
Statistical Analysis 1: Comparison: Placebo + LenDex vs Ixazomib + LenDex; Test type: Superiority; p = 0.9195, Regression, Logistic; Logistic regression model with prognostic factor: age (<75 years vs >=75) and ISS (stage I or II vs stage III); Odds Ratio (OR) = 0.980, 95% CI 2-sided [0.656 to 1.463] — Odds ratio > 1 favors Ixazomib+LenDex versus LenDex alone

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved CR + partial response (PR) + very good partial response (VGPR) (including sCR) or better relative to the ITT population during treatment period. CR was defined as negative immunofixation of serum and urine along with the disappearance of any soft tissue plasmacytomas and <5 % PC's in bone marrow. PR was defined as ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% along with ≥50% reduction in the size of soft tissue plasmacytomas. VGPR was defined as ≥90% in serum M-component plus urine M-component <100 mg/24. sCR is defined as stringent complete response. Percentages are rounded off to nearest whole numbers.
Time Frame: Up to approximately 9 years
Population: ITT population included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 354 | 351
percentage of participants | 80 | 82
Statistical Analysis 1: Comparison: Placebo + LenDex vs Ixazomib + LenDex; Test type: Superiority; p = 0.436, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.79 to 1.70] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from the date of randomization to the first documentation of PR or better, as measured by IMWG criteria.
Time Frame: Up to approximately 9 years
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 354 | 351
months | 1.87 [1.15 to 1.87] | 1.02 [0.99 to 1.08]
Statistical Analysis 1: Comparison: Placebo + LenDex vs Ixazomib + LenDex; Test type: Superiority; p < 0.001, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.402, 95% CI 2-sided [1.185 to 1.659] — Hazard ratio is based on an unadjusted Cox's proportional hazard regression model stratified by age (<75 years vs >=75), ISS (stage I or II vs stage III), and BPI-SF worst pain score (<4 vs >=4) at screening

7. Secondary Outcome: Duration of Response
Description: Duration of response was measured as the time from the date of first documentation of PR or better to the date of first documented progression (PD) for responders, as measured by IMWG criteria.
Time Frame: Up to approximately 9 years
Population: Response-evaluable population was defined as all participants in the ITT population who receive at least 1 dose of any study drug, have measurable disease at baseline, and at least 1 post baseline response assessment assessed by an IRC. Overall number of participants analyzed are the number of responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 281 | 287
months | 37.5 [25.69 to 50.27] | 50.6 [39.98 to NA] — Upper limit of CI was not estimable as participants without documentation of PD at the date of last response assessment that is stable disease (SD) or better were censored.

8. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression was defined as the time from randomization to the date of first documented disease progression.
Time Frame: Up to approximately 9 years
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 354 | 351
months | 26.8 [21.22 to 37.91] | 45.8 [31.84 to 56.25]
Statistical Analysis 1: Comparison: Placebo + LenDex vs Ixazomib + LenDex; Test type: Superiority; p = 0.008, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.738, 95% CI 2-sided [0.589 to 0.925] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Progression Free Survival (PFS)-2
Description: PFS2 was defined as the time from the date of randomization to the date of documentation of disease progression on the subsequent line of anticancer therapy, as assessed by the investigator in accordance with IMWG criteria, or death due to any cause, whichever occurs first.
Time Frame: Up to approximately 9 years
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 354 | 351
months | 52.2 [45.21 to 61.90] | 63.2 [54.70 to NA] — Upper limit of CI was not estimable to due insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo + LenDex vs Ixazomib + LenDex; Test type: Superiority; p = 0.189, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.859, 95% CI 2-sided [0.684 to 1.078] — [estimate comment as in outcome 6, analysis 1]

10. Secondary Outcome: Number of Participants With Shifts From Baseline to Worst Value in Eastern Cooperative Oncology Group (ECOG) Performance Score
Description: Eastern Cooperative Oncology Group (ECOG) scale score ranged from 0 to 5, where 0 indicated normal activity and 5 indicated death. The data is reported for those categories where at least 1 participant had worst post-baseline value for each ECOG score.
Time Frame: Up to approximately 9 years
Population: Safety population is defined as all participants who receive at least 1 dose of any study drug. Overall number of participants analyzed indicates number of participants available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 344 | 340
Participants
  Baseline Score 0, Post-Baseline Score 0 | 23 | 23
  Baseline Score 0, Post-Baseline Score 1 | 57 | 52
  Baseline Score 0, Post-Baseline Score 2 | 20 | 23
  Baseline Score 0, Post-Baseline Score 3 | 2 | 10
  Baseline Score 1, Post-Baseline Score 0 | 1 | 1
  Baseline Score 1, Post-Baseline Score 1 | 96 | 104
  Baseline Score 1, Post-Baseline Score 2 | 72 | 57
  Baseline Score 1, Post-Baseline Score 3 | 18 | 9
  Baseline Score 1, Post-Baseline Score 4 | 6 | 4
  Baseline Score 2, Post-Baseline Score 1 | 12 | 8
  Baseline Score 2, Post-Baseline Score 2 | 28 | 35
  Baseline Score 2, Post-Baseline Score 3 | 7 | 11
  Baseline Score 2, Post-Baseline Score 4 | 2 | 3

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant administered a medicinal investigational drug. The untoward medical occurrence does not necessarily have to have a causal relationship with treatment. An SAE is any untoward medical occurrence that results in death; is life-threatening; requires inpatient hospitalization or prolongation of present hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect or is a medically important event that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the participant or may require intervention to prevent one of other outcomes listed in definition above, or involves suspected transmission via a medicinal product of an infectious agent.
Time Frame: From the date of randomization through 30 days after the last dose of study drug up to end of study (up to approximately 9 years)
Population: Safety population is defined as all participants who receive at least 1 dose of any study drug. Data for safety is summarized as per the duration of exposure to study treatment (exposure up to 18 cycles; exposure ≥19 cycles).
Measure: Count of Participants; unit: Participants
Groups:
- Placebo + LenDex (Exposure Up to 18 Cycles): Participants who were randomly assigned to receive placebo matching capsule single oral dose on Days 1, 8 and 15 along with standard regimen of LenDex (lenalidomide 25 mg capsules orally on Days 1-21 and dexamethasone 40 mg tablets orally on Days 1, 8, 15 and 22) up to 18 cycles (each cycle was of 28 days).
- Ixazomib+ LenDex (Exposure Up to 18 Cycles): Participants who were randomly assigned to receive Ixazomib 4.0 mg capsule single oral dose on Days 1, 8 and 15 along with standard regimen of LenDex (lenalidomide 25 mg capsules orally on Days 1-21 and dexamethasone 40 mg tablets orally on Days 1, 8, 15 and 22) up to 18 cycles (each cycle was of 28 days).
- Placebo + LenDex (Exposure ≥19 Cycles): Participants who were randomly assigned to receive placebo matching capsule single oral dose on Days 1, 8 and 15 along with standard regimen of LenDex (lenalidomide 25 mg capsules orally on Days 1-21 and dexamethasone 40 mg tablets orally on Days 1, 8, 15 and 22) up to 18 cycles (each cycle was of 28 days). Following Cycle 18, participants received 3.0 mg ixazomib placebo matching capsule as single oral dose on Days 1, 8 and 15 along with lenalidomide 10 mg capsules orally on Days 1-21 in each 28-day cycle until progressive disease or unacceptable toxicity, whichever comes first up to end of study (up to approximately 109 months).
- Ixazomib + LenDex (Exposure ≥19 Cycles): Participants who were randomly assigned to receive Ixazomib 4.0 mg placebo matching capsule single oral dose on Days 1, 8 and 15 along with standard regimen of LenDex (lenalidomide 25 mg capsules orally on Days 1-21 and dexamethasone 40 mg tablets orally on Days 1, 8, 15 and 22) up to 18 cycles (each cycle was of 28 days). Following Cycle 18, participants received 3.0 mg ixazomib capsule as single oral dose on Days 1, 8 and 15 along with lenalidomide 10 mg capsules orally on Days 1-21 in each 28-day cycle until progressive disease or unacceptable toxicity, whichever comes first up to end of study (up to approximately 109 months).
Arm/Group | Placebo + LenDex (Exposure Up to 18 Cycles) | Ixazomib+ LenDex (Exposure Up to 18 Cycles) | Placebo + LenDex (Exposure ≥19 Cycles) | Ixazomib + LenDex (Exposure ≥19 Cycles)
Number analyzed (Participants) | 160 | 163 | 189 | 191
Participants
  TEAEs | 160 | 163 | 189 | 191
  SAEs | 105 | 119 | 119 | 125

12. Secondary Outcome: Number of Participants With Abnormal Serum Chemistry and Hematology Laboratory Values Based on Treatment-emergent Adverse Events (TEAEs)
Description: The laboratory values assessment included serum chemistry and hematology. The Serum chemistry assessment included blood urea nitrogen (BUN), creatinine, bilirubin (total), urate, lactate dehydrogenase, phosphate, albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), glucose, sodium, potassium, calcium, chloride, carbon dioxide (CO2), magnesium, thyroid stimulating hormone (TSH). Hematology assessment included hemoglobin, hematocrit, platelet (count), leukocytes with differential neutrophils (ANC). Participants with abnormal serum chemistry laboratory values reported as TEAEs are reported. TEAEs were defined as events that occurred after administration of the first dose of any agent in the study drug regimen and through 30 days after the last dose of any agent in the study drug regimen.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + LenDex (Exposure Up to 18 Cycles) | Ixazomib+ LenDex (Exposure Up to 18 Cycles) | Placebo + LenDex (Exposure ≥19 Cycles) | Ixazomib + LenDex (Exposure ≥19 Cycles)
Number analyzed (Participants) | 160 | 163 | 189 | 191
Participants
  Hypokalaemia | 16 | 33 | 33 | 39
  Blood creatinine increased | 9 | 6 | 12 | 16
  Hypophosphataemia | 2 | 9 | 3 | 9
  Hypomagnesaemia | 8 | 6 | 11 | 15
  Hyponatraemia | 7 | 10 | 8 | 7
  Hyperglycaemia | 4 | 7 | 16 | 6
  Hypocalcaemia | 13 | 6 | 12 | 4
  Hyperkalaemia | 3 | 7 | 3 | 3
  Alanine aminotransferase increased | 1 | 1 | 4 | 10
  Iron deficiency | 2 | 1 | 2 | 7
  Hypercalcaemia | 6 | 2 | 1 | 5
  Creatinine renal clearance decreased | 2 | 1 | 7 | 4
  Hypoalbuminaemia | 5 | 2 | 1 | 3
  Aspartate aminotransferase increased | 1 | 0 | 3 | 5
  Hyperuricaemia | 2 | 2 | 1 | 2
  Anaemia | 57 | 53 | 52 | 58
  Thrombocytopenia | 15 | 34 | 14 | 24
  Neutropenia | 36 | 15 | 48 | 39
  Neutrophil count decreased | 11 | 5 | 13 | 18
  Platelet count decreased | 6 | 6 | 4 | 15
  Lymphopenia | 0 | 7 | 2 | 4
  Febrile neutropenia | 5 | 7 | 2 | 2
  Leukopenia | 3 | 6 | 4 | 2
  International normalised ratio increased | 1 | 4 | 0 | 4
  Pancytopenia | 2 | 3 | 1 | 2
  Iron deficiency anaemia | 1 | 1 | 1 | 4
  White blood cell count decreased | 5 | 1 | 3 | 2
  Lymphocyte count decreased | 1 | 2 | 3 | 0

13. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQOL) Measured by European Organisation for Research and Treatment of Cancer-Quality of Life Questionnaire (EORTC-QLQ)-C30 Scale Total Score
Description: EORTC-QLQ-C30 scale was used to assess HRQOL in cancer participants and contains 30 items. Subscale with individual items include physical functioning items 1-5, role functioning items 6-7, emotional functioning items 21-24, cognitive functioning items 20, 25, social functioning items 26-27, quality of life items 29-30, fatigue items 10, 12, 18, nausea and vomiting items 14-15, pain items 9, 19, dyspnoea item 8, insomnia item 11, appetite loss item 13, constipation item 16, diarrhoea item 17, financial difficulties item 28. Raw scores were converted into scale scores ranging from 0 to 100. For the functional scales and the global health status scale, higher scores represent better HRQOL; whereas for the symptom scales lower scores represent better HRQOL. Positive change in functional and global health status scale indicated improvement; negative change for the symptom scales indicates improvement.
Time Frame: Baseline to approximately 9 years
Population: ITT population included all participants who were randomized. Overall number of participants analyzed is the number of participants available for analyses. Number analyzed indicates the number of participants available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 353 | 351
score on a scale
  Global Health Status/QoL: Baseline: number analyzed (Participants) | 352 | 351
  Global Health Status/QoL: Baseline | 55.2 (23.53) | 56.4 (23.66)
  Global Health Status/QoL: End of Treatment: number analyzed (Participants) | 220 | 217
  Global Health Status/QoL: End of Treatment | -2.2 (26.03) | -4.1 (29.48)
  Physical Functioning: Baseline: number analyzed (Participants) | 353 | 350
  Physical Functioning: Baseline | 60.0 (28.73) | 61.4 (27.96)
  Physical Functioning: End of Treatment: number analyzed (Participants) | 223 | 217
  Physical Functioning: End of Treatment | 1.7 (26.81) | 0.3 (28.23)
  Role Functioning: Baseline: number analyzed (Participants) | 352 | 350
  Role Functioning: Baseline | 54.9 (36.52) | 56.5 (36.60)
  Role Functioning: End of Treatment: number analyzed (Participants) | 223 | 217
  Role Functioning: End of Treatment | -0.3 (36.25) | -1.8 (36.74)
  Emotional Functioning: Baseline | 73.5 (23.09) | 72.6 (24.84)
  Emotional Functioning: End of Treatment: number analyzed (Participants) | 222 | 217
  Emotional Functioning: End of Treatment | -2.4 (21.70) | -0.5 (24.35)
  Cognitive Functioning: Baseline | 77.8 (22.97) | 78.3 (25.92)
  Cognitive Functioning: End of Treatment: number analyzed (Participants) | 222 | 217
  Cognitive Functioning: End of Treatment | -3.2 (25.14) | -5.1 (24.70)
  Social Functioning: Baseline: number analyzed (Participants) | 351 | 351
  Social Functioning: Baseline | 69.1 (32.54) | 69.5 (33.01)
  Social Functioning: End of Treatment: number analyzed (Participants) | 220 | 217
  Social Functioning: End of Treatment | -2.9 (31.56) | -2.5 (36.57)
  Fatigue: Baseline: number analyzed (Participants) | 353 | 350
  Fatigue: Baseline | 44.6 (28.30) | 40.8 (27.69)
  Fatigue: End of Treatment: number analyzed (Participants) | 223 | 218
  Fatigue: End of Treatment | -2.3 (27.75) | 4.5 (31.04)
  Pain: Baseline | 45.6 (34.04) | 42.5 (33.51)
  Pain: End of Treatment: number analyzed (Participants) | 225 | 218
  Pain: End of Treatment | -5.5 (33.77) | -3.5 (34.55)
  Nausea and Vomiting: Baseline: number analyzed (Participants) | 353 | 350
  Nausea and Vomiting: Baseline | 7.1 (15.75) | 8.1 (18.49)
  Nausea and Vomiting: End of Treatment: number analyzed (Participants) | 224 | 218
  Nausea and Vomiting: End of Treatment | -0.5 (19.80) | 1.6 (25.22)
  Dyspnoea: Baseline: number analyzed (Participants) | 352 | 350
  Dyspnoea: Baseline | 26.2 (30.25) | 24.0 (29.35)
  Dyspnoea: End of Treatment: number analyzed (Participants) | 222 | 217
  Dyspnoea: End of Treatment | -3.6 (30.86) | 2.8 (33.83)
  Insomnia: Baseline: number analyzed (Participants) | 353 | 350
  Insomnia: Baseline | 30.3 (30.31) | 34.3 (32.20)
  Insomnia: End of Treatment: number analyzed (Participants) | 223 | 217
  Insomnia: End of Treatment | -1.5 (35.06) | -1.1 (36.06)
  Appetite Loss: Baseline: number analyzed (Participants) | 353 | 350
  Appetite Loss: Baseline | 25.4 (33.14) | 25.5 (33.04)
  Appetite Loss: End of Treatment: number analyzed (Participants) | 223 | 218
  Appetite Loss: End of Treatment | -1.2 (37.42) | 3.4 (38.65)
  Constipation: Baseline: number analyzed (Participants) | 352 | 351
  Constipation: Baseline | 25.9 (32.94) | 24.9 (32.19)
  Constipation: End of Treatment: number analyzed (Participants) | 222 | 218
  Constipation: End of Treatment | -7.1 (39.03) | -5.7 (35.83)
  Diarrhoea: Baseline: number analyzed (Participants) | 352 | 351
  Diarrhoea: Baseline | 8.2 (19.45) | 6.7 (16.58)
  Diarrhoea: End of Treatment: number analyzed (Participants) | 221 | 217
  Diarrhoea: End of Treatment | 10.7 (27.72) | 18.3 (31.73)
  Financial Difficulties: Baseline: number analyzed (Participants) | 352 | 351
  Financial Difficulties: Baseline | 12.5 (24.04) | 12.3 (24.03)
  Financial Difficulties: End of Treatment: number analyzed (Participants) | 220 | 216
  Financial Difficulties: End of Treatment | 2.0 (27.42) | 0.8 (25.61)

14. Secondary Outcome: Change From Baseline in HRQOL Measured by EORTC-QLQ-MY20 Scale
Description: EORTC QLQ-MY20 was a validated questionnaire to assess the overall quality of life in participants with multiple myeloma. The scale has 20 questions. Subscale and individual items include future perspective items 18-20, body image item 17, disease symptoms items 1-6, side effects of treatment items 7-16. Raw scores are averaged, and transformed to 0-100 scale, where higher score is better quality of life. Positive change indicates improvement.
Time Frame: Baseline to approximately 9 years
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 352 | 350
score on a scale
  Disease Symptoms: Baseline | 30.3 (23.76) | 29.2 (22.97)
  Disease Symptoms: End of Treatment: number analyzed (Participants) | 222 | 215
  Disease Symptoms: End of Treatment | -3.1 (20.74) | -5.3 (22.44)
  Side-Effects: Baseline | 18.0 (14.53) | 17.6 (15.04)
  Side-Effects: End of Treatment: number analyzed (Participants) | 222 | 214
  Side-Effects: End of Treatment | 1.7 (14.52) | 3.3 (15.91)
  Body Image: Baseline: number analyzed (Participants) | 346 | 346
  Body Image: Baseline | 81.7 (27.67) | 81.2 (29.11)
  Body Image: End of Treatment: number analyzed (Participants) | 215 | 207
  Body Image: End of Treatment | -7.8 (31.93) | -2.3 (29.66)
  Future Perspective: Baseline: number analyzed (Participants) | 350 | 349
  Future Perspective: Baseline | 57.3 (25.95) | 55.0 (28.47)
  Future Perspective: End of Treatment: number analyzed (Participants) | 220 | 211
  Future Perspective: End of Treatment | 4.4 (24.85) | 6.0 (25.69)

15. Secondary Outcome: OS in High-risk Population Carrying Del(17p), t(4;14), or t(14;16) Mutations
Description: OS was defined as the time from the date of randomization to the date of death, as assessed in high-risk population carrying del(17p), t(4;14), or t(14;16) mutations. High risk category includes t(4;14), t(14;16), or del(17) abnormalities.
Time Frame: From the date of randomization to death due to any cause (Up to approximately 9 years)
Population: ITT population included all participants who were randomized. Overall number of participants analyzed indicates the number of participants from the high-risk category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 63 | 60
months | 43.1 [33.84 to 57.82] | 39.0 [25.43 to NA] — Upper range of CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo + LenDex vs Ixazomib + LenDex; OS in High-risk Population Carrying Del(17p), Amp(1q21), t(4;14), or t(14;16) Mutations; Test type: Superiority; p = 0.662, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.118, 95% CI 2-sided [0.678 to 1.845] — [estimate comment as in outcome 6, analysis 1]

16. Secondary Outcome: PFS in High-risk Population Carrying Del(17p), t(4;14), or t(14;16) Mutations
Description: PFS was defined as the time from the date of randomization to the date of first documentation of progressive disease based on central laboratory results and IMWG criteria as evaluated by an independent review committee (IRC) or death due to any cause, whichever occurs first, as assessed in high-risk population carrying del(17p), t(4;14), or t(14;16) mutations.
Time Frame: Up to approximately 9 years
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 63 | 60
months | 17.5 [12.12 to 20.30] | 22.4 [12.16 to 42.84]
Statistical Analysis 1: Comparison: Placebo + LenDex vs Ixazomib + LenDex; PFS in High-risk Population Carrying del(17p), t(4;14), or t(14;16) Mutations; Test type: Superiority; p = 0.271, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.760, 95% CI 2-sided [0.466 to 1.240] — [estimate comment as in outcome 6, analysis 1]

17. Secondary Outcome: Percentage of Participants With MRD-Negative Status as Assessed by Flow Cytometry
Description: The absence of minimal residual disease (MRD negativity) was tested in all participants who achieve a CR and maintained it until Cycle 18, using bone marrow aspirates.
Time Frame: Up to Cycle 18 (cycle length = 28 days)
Population: Response-evaluable population includes all participants in the ITT population who receive at least 1 dose of any study drug, have measurable disease at baseline, and at least 1 post baseline response assessment assessed by an IRC. Percentages are rounded off to the nearest single decimal.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 347 | 335
percentage of participants | 50 | 59

18. Secondary Outcome: Time to Pain Progression
Description: Time to pain progression was assessed as the time from randomization to the date of initial progression classification. Pain progression was defined as the occurrence of 1 of the following and confirmed by 2 consecutive evaluations (To qualify as progression, the participant must have a BPI-SF worst pain score > 4 during pain progression): 1) a ≥ 2 point and 30% increase from Baseline in BPI-SF worst pain score without an increase in analgesic use, or 2) a 25% or more increase in analgesic use from Baseline without a decrease in BPI-SF worst pain score from Baseline. Brief Pain Inventory - Short Form (m-BPI-SF) is a participant rated 11-point Likert rating scale ranged from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: Up to approximately 9 years
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + LenDex | Ixazomib + LenDex
Number analyzed (Participants) | 354 | 351
months | 47.1 [30.88 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events. | NA [57.59 to NA] — Median and upper limit of CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo + LenDex vs Ixazomib + LenDex; Time to Pain Progression; Test type: Superiority; p = 0.260, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.860, 95% CI 2-sided [0.661 to 1.120] — [estimate comment as in outcome 6, analysis 1]

19. Secondary Outcome: Cmax: Maximum Plasma Concentration for Ixazomib
Time Frame: Cycle 1 Day 1: Post-dose at multiple timepoints up to 4 hours; Pre-dose at Cycle 1 Day 14, Cycles 2-3 Day 1 and Day 14, Cycles 4-11 Day 1 (Each cycle length = 28 days)
Population: Pharmacokinetic (PK) analysis population is defined as subjects with at least one PK sample that was collected and analyzed. Overall number of participants analyzed is the number of participants available for analyses. Number analyzed indicates the number of participants available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Groups:
- Ixazomib: Participants who were randomly assigned to receive Ixazomib 4.0 mg capsules orally once on Days 1,8,15 and lenalidomide 25 mg capsules orally on days 1-21 and dexamethasone 40 mg tablets orally on Days 1,8, 15 and 22, during every 28-day cycle for the first 18 cycles.
  After Cycle 18 dexamethasone was discontinued and participants continued to receive ixazomib capsule and lenalidomide at reduced doses until progressive disease or unacceptable toxicity, whichever comes first, up to end of study (up to approximately 109 months).
Arm/Group | Ixazomib
Number analyzed (Participants) | 331
nanograms per milliliter
  Cycle 1 Day 1: 1 Hour Post-dose | 44.745 (35.9404)
  Cycle 1 Day 1: 4 Hours Post-dose: number analyzed (Participants) | 320
  Cycle 1 Day 1: 4 Hours Post-dose | 16.253 (17.0407)
  Cycle 1 Day 14: Pre-dose: number analyzed (Participants) | 327
  Cycle 1 Day 14: Pre-dose | 7.867 (15.4420)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 320
  Cycle 2 Day 1: Pre-dose | 2.664 (2.2770)
  Cycle 2 Day 14: Pre-dose: number analyzed (Participants) | 302
  Cycle 2 Day 14: Pre-dose | 8.521 (14.7411)
  Cycle 3 Day 1: Pre-dose: number analyzed (Participants) | 300
  Cycle 3 Day 1: Pre-dose | 2.763 (1.6318)
  Cycle 3 Day 14: Pre-dose: number analyzed (Participants) | 275
  Cycle 3 Day 14: Pre-dose | 8.490 (17.6720)
  Cycle 4 Day 1: Pre-dose: number analyzed (Participants) | 284
  Cycle 4 Day 1: Pre-dose | 3.284 (6.1116)
  Cycle 5 Day 1: Pre-dose: number analyzed (Participants) | 270
  Cycle 5 Day 1: Pre-dose | 3.594 (13.2046)
  Cycle 6 Day 1: Pre-dose: number analyzed (Participants) | 260
  Cycle 6 Day 1: Pre-dose | 2.603 (1.5242)
  Cycle 7 Day 1: Pre-dose: number analyzed (Participants) | 258
  Cycle 7 Day 1: Pre-dose | 2.598 (1.4658)
  Cycle 8 Day 1: Pre-dose: number analyzed (Participants) | 251
  Cycle 8 Day 1: Pre-dose | 2.539 (1.5549)
  Cycle 9 Day 1: Pre-dose: number analyzed (Participants) | 242
  Cycle 9 Day 1: Pre-dose | 2.593 (2.0867)
  Cycle 10 Day 1: Pre-dose: number analyzed (Participants) | 238
  Cycle 10 Day 1: Pre-dose | 2.536 (1.7431)
  Cycle 11 Day 1: Pre-dose: number analyzed (Participants) | 224
  Cycle 11 Day 1: Pre-dose | 2.667 (4.5448)
  Cycle 12 Day 1: Pre-dose: number analyzed (Participants) | 217
  Cycle 12 Day 1: Pre-dose | 2.686 (1.8949)

20. Secondary Outcome: Percentage of Participants With New or Worsening of Existing Skeletal-related Events (SREs)
Description: SRE is defined as new fractures [including vertebral compression fractures], irradiation of or surgery on bone, or spinal cord compression.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Number; unit: percentage of partcipants
Arm/Group | Placebo + LenDex (Exposure Up to 18 Cycles) | Ixazomib+ LenDex (Exposure Up to 18 Cycles) | Placebo + LenDex (Exposure ≥19 Cycles) | Ixazomib + LenDex (Exposure ≥19 Cycles)
Number analyzed (Participants) | 160 | 163 | 189 | 191
percentage of partcipants | 14 | 10 | 28 | 25

ADVERSE EVENTS:
Time Frame: From the date of randomization through 30 days after the last dose of study drug up to end of study (up to approximately 9 years)
Description: Safety population included all participants who received at least 1 dose of any drug. 4 participants who were randomized to the placebo received ixazomib during the study and were included in the ixazomib arm for the safety population. 1 participant randomized to each arm withdrew from the study and were not included in the safety population. Data for safety is summarized as per the duration of exposure to study treatment (exposure up to 18 cycles; exposure ≥19 cycles).
Arm/Group | Placebo + LenDex (Exposure Up to 18 Cycles) | Ixazomib+ LenDex (Exposure Up to 18 Cycles) | Placebo + LenDex (Exposure ≥19 Cycles) | Ixazomib + LenDex (Exposure ≥19 Cycles)
All-Cause Mortality (participants affected / at risk) | 107/160 | 95/163 | 63/189 | 63/191
Serious Adverse Events (participants affected / at risk) | 105/160 | 119/163 | 119/189 | 125/191
Other Adverse Events (participants affected / at risk) | 159/160 | 162/163 | 189/189 | 191/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + LenDex (Exposure Up to 18 Cycles) (N=160) | Ixazomib+ LenDex (Exposure Up to 18 Cycles) (N=163) | Placebo + LenDex (Exposure ≥19 Cycles) (N=189) | Ixazomib + LenDex (Exposure ≥19 Cycles) (N=191)
Pneumonia (Infections and infestations) | 16 | 22 | 13 | 22
Bronchitis (Infections and infestations) | 0 | 3 | 5 | 4
Lower respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pleural infection (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 4 | 4 | 4 | 1
Septic shock (Infections and infestations) | 4 | 4 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 3 | 6
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 2 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 2
Cystitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Superinfection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 4 | 2 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 2 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 3 | 1 | 0
Toxic shock syndrome staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 1 | 3 | 2
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 3
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral uveitis (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 1
Abscess jaw (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis aspergillus (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Prostatitis Escherichia coli (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 1 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Bartholinitis (Infections and infestations) | 0 | 0 | 1 | 0
Fungal oesophagitis (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis E (Infections and infestations) | 1 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 6 | 12
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4 | 5
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 1 | 0
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 4
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Sarcomatoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 8 | 1 | 7
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric volvulus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 5 | 5 | 2 | 3
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 3 | 3 | 4
Sudden death (General disorders) | 1 | 1 | 0 | 3
Death (General disorders) | 1 | 1 | 0 | 1
Asthenia (General disorders) | 2 | 1 | 1 | 1
Malaise (General disorders) | 0 | 1 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 1
Pain (General disorders) | 1 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 1 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 1 | 0 | 0
Stent-graft endoleak (General disorders) | 0 | 0 | 0 | 1
Hyperthermia (General disorders) | 1 | 0 | 0 | 0
Complication associated with device (General disorders) | 0 | 0 | 1 | 0
Incarcerated hernia (General disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 1 | 3
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Thalamic infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Thalamus haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 4 | 6 | 14
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 2
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 27 | 23 | 57 | 85
Spinal claudication (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 3 | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 5 | 1 | 2 | 3
Atrial fibrillation (Cardiac disorders) | 3 | 3 | 3 | 4
Supraventricular tachycardia (Cardiac disorders) | 2 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 2 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 3 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 2 | 3
Cardiac arrest (Cardiac disorders) | 0 | 4 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 5 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 5 | 7 | 20 | 10
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 4
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 4 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Aortic injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 11 | 10 | 5 | 12
Decreased appetite (Metabolism and nutrition disorders) | 45 | 34 | 35 | 45
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 3
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 8 | 5 | 2 | 3
Renal failure (Renal and urinary disorders) | 3 | 1 | 0 | 2
Renal impairment (Renal and urinary disorders) | 1 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 5 | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 2 | 5 | 4
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 2 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 2 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 5 | 2
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0
Obsessive thoughts (Psychiatric disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 2 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Staphylococcus test positive (Investigations) | 1 | 0 | 0 | 0
Blast cells present (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Optic nerve sheath haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Amaurosis (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 3 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Testicular oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Device breakage (Product Issues) | 0 | 0 | 0 | 1
Device loosening (Product Issues) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural Heamatoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Acute erythroid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Myeloma cast nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0
Senile dementia (Nervous system disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Prosthetic cardiac valve malfunction (Product Issues) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + LenDex (Exposure Up to 18 Cycles) (N=160) | Ixazomib+ LenDex (Exposure Up to 18 Cycles) (N=163) | Placebo + LenDex (Exposure ≥19 Cycles) (N=189) | Ixazomib + LenDex (Exposure ≥19 Cycles) (N=191)
Oedema peripheral (General disorders) | 52 | 66 | 64 | 106
Fatigue (General disorders) | 53 | 41 | 52 | 69
Asthenia (General disorders) | 44 | 36 | 53 | 58
Pyrexia (General disorders) | 20 | 30 | 29 | 33
Peripheral swelling (General disorders) | 8 | 8 | 12 | 17
Malaise (General disorders) | 3 | 6 | 16 | 17
Influenza like illness (General disorders) | 4 | 1 | 11 | 16
Non-cardiac chest pain (General disorders) | 2 | 4 | 10 | 14
Chills (General disorders) | 10 | 11 | 7 | 12
Diarrhoea (Gastrointestinal disorders) | 48 | 68 | 115 | 147
Constipation (Gastrointestinal disorders) | 61 | 59 | 82 | 92
Nausea (Gastrointestinal disorders) | 35 | 55 | 63 | 78
Vomiting (Gastrointestinal disorders) | 13 | 41 | 33 | 66
Dry mouth (Gastrointestinal disorders) | 14 | 11 | 12 | 13
Stomatitis (Gastrointestinal disorders) | 9 | 10 | 8 | 15
Abdominal pain upper (Gastrointestinal disorders) | 13 | 8 | 29 | 23
Abdominal pain (Gastrointestinal disorders) | 10 | 7 | 38 | 30
Dyspepsia (Gastrointestinal disorders) | 16 | 5 | 22 | 21
Haemorrhoids (Gastrointestinal disorders) | 6 | 1 | 15 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 4 | 10 | 13
Abdominal distension (Gastrointestinal disorders) | 6 | 1 | 11 | 11
Toothache (Gastrointestinal disorders) | 4 | 3 | 15 | 8
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 10 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 | 37 | 22 | 43
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 16 | 29 | 37
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 11 | 22 | 31
Rash macular (Skin and subcutaneous tissue disorders) | 3 | 11 | 11 | 27
Erythema (Skin and subcutaneous tissue disorders) | 2 | 11 | 20 | 16
Rash (Skin and subcutaneous tissue disorders) | 9 | 11 | 7 | 18
Night sweats (Skin and subcutaneous tissue disorders) | 9 | 9 | 9 | 5
Rash papular (Skin and subcutaneous tissue disorders) | 8 | 8 | 4 | 12
Rash erythematous (Skin and subcutaneous tissue disorders) | 10 | 6 | 3 | 18
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3 | 8 | 13
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 5 | 10
Dizziness (Nervous system disorders) | 31 | 27 | 36 | 31
Peripheral sensory neuropathy (Nervous system disorders) | 27 | 23 | 57 | 83
Headache (Nervous system disorders) | 22 | 15 | 36 | 33
Tremor (Nervous system disorders) | 23 | 14 | 27 | 19
Dysgeusia (Nervous system disorders) | 14 | 9 | 12 | 32
Paraesthesia (Nervous system disorders) | 13 | 9 | 21 | 25
Hypoaesthesia (Nervous system disorders) | 7 | 6 | 11 | 14
Sciatica (Nervous system disorders) | 3 | 4 | 11 | 16
Neuropathy peripheral (Nervous system disorders) | 3 | 2 | 9 | 14
Syncope (Nervous system disorders) | 0 | 0 | 6 | 13
Urinary tract infection (Infections and infestations) | 14 | 19 | 27 | 30
Bronchitis (Infections and infestations) | 13 | 13 | 51 | 74
Nasopharyngitis (Infections and infestations) | 13 | 13 | 71 | 62
Upper respiratory tract infection (Infections and infestations) | 17 | 10 | 47 | 48
Herpes zoster (Infections and infestations) | 4 | 4 | 4 | 24
Rhinitis (Infections and infestations) | 5 | 2 | 21 | 23
Pneumonia (Infections and infestations) | 6 | 7 | 20 | 24
Sinusitis (Infections and infestations) | 1 | 5 | 6 | 18
Conjunctivitis (Infections and infestations) | 2 | 2 | 5 | 18
Gastroenteritis (Infections and infestations) | 4 | 4 | 15 | 15
Influenza (Infections and infestations) | 3 | 3 | 22 | 13
Cystitis (Infections and infestations) | 2 | 2 | 12 | 13
Cellulitis (Infections and infestations) | 5 | 2 | 3 | 11
Pharyngitis (Infections and infestations) | 1 | 2 | 10 | 10
Tooth infection (Infections and infestations) | 2 | 2 | 11 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 26 | 67 | 64
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 | 18 | 50 | 50
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 23 | 81 | 76
Muscle spasms (Musculoskeletal and connective tissue disorders) | 27 | 15 | 50 | 52
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 | 12 | 27 | 25
Muscular weakness (Musculoskeletal and connective tissue disorders) | 12 | 9 | 19 | 18
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 14 | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 7 | 25 | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 5 | 24 | 33
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 4 | 24 | 20
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 13 | 24
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 16
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 7 | 11 | 12
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 20 | 9
Decreased appetite (Metabolism and nutrition disorders) | 45 | 34 | 34 | 45
Hypokalaemia (Metabolism and nutrition disorders) | 16 | 33 | 33 | 39
Dehydration (Metabolism and nutrition disorders) | 11 | 10 | 5 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 10 | 7 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 9 | 3 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 13 | 6 | 12 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 6 | 11 | 15
Gout (Metabolism and nutrition disorders) | 4 | 1 | 14 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 7 | 15 | 6
Anaemia (Blood and lymphatic system disorders) | 56 | 51 | 51 | 58
Thrombocytopenia (Blood and lymphatic system disorders) | 15 | 32 | 14 | 24
Neutropenia (Blood and lymphatic system disorders) | 36 | 15 | 48 | 39
Insomnia (Psychiatric disorders) | 27 | 30 | 68 | 70
Anxiety (Psychiatric disorders) | 15 | 22 | 25 | 26
Depression (Psychiatric disorders) | 10 | 18 | 14 | 26
Confusional state (Psychiatric disorders) | 15 | 16 | 11 | 11
Agitation (Psychiatric disorders) | 3 | 4 | 10 | 11
Irritability (Psychiatric disorders) | 3 | 1 | 11 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 28 | 37 | 53
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 | 21 | 26 | 39
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 7 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 7 | 16 | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 14 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 12 | 12
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 5 | 12
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 10 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 12 | 4
Weight decreased (Investigations) | 20 | 24 | 30 | 35
Neutrophil count decreased (Investigations) | 11 | 5 | 13 | 18
Blood creatinine increased (Investigations) | 8 | 6 | 12 | 16
Platelet count decreased (Investigations) | 6 | 6 | 4 | 15
Hypertension (Vascular disorders) | 9 | 6 | 18 | 29
Hypotension (Vascular disorders) | 12 | 17 | 11 | 15
Haematoma (Vascular disorders) | 1 | 2 | 7 | 10
Flushing (Vascular disorders) | 5 | 4 | 12 | 6
Hot flush (Vascular disorders) | 2 | 0 | 14 | 4
Deep vein thrombosis (Vascular disorders) | 15 | 5 | 13 | 4
Cardiac failure (Cardiac disorders) | 3 | 9 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 8 | 6 | 11 | 6
Palpitations (Cardiac disorders) | 0 | 0 | 8 | 11
Fall (Injury, poisoning and procedural complications) | 9 | 8 | 35 | 45
Contusion (Injury, poisoning and procedural complications) | 7 | 3 | 20 | 19
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 11 | 6
Cataract (Eye disorders) | 6 | 1 | 41 | 54
Vision blurred (Eye disorders) | 6 | 6 | 22 | 25
Dry eye (Eye disorders) | 1 | 5 | 6 | 17
Vertigo (Ear and labyrinth disorders) | 4 | 3 | 18 | 22
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 6 | 10
Dental caries (Gastrointestinal disorders) | 2 | 0 | 11 | 6
Alanine aminotransferase increased (Investigations) | 1 | 1 | 4 | 10
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 5 | 8 | 10
Skin laceration (Injury, poisoning and procedural complications) | 4 | 2 | 10 | 8
Memory impairment (Nervous system disorders) | 3 | 4 | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT01850524/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT01850524/SAP_001.pdf